CLINICAL TRIAL: NCT01660191
Title: A Study Comparing the Effects of Pitavastatin, Atorvastatin, and Rosuvastatin on Plasma Levels of CoQ10 (SPARQ)
Brief Title: A Study Comparing CoQ10 Levels While Taking 3 Different Statins
Acronym: SPARQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Kowa Pharmaceuticals America, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Patrick Moriarty, MD, FACP, FACC, Director, Atherosclerosis & LDL-Apheresis Center, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12943
Record Dates: First submitted 2012-05-21; First posted 2012-08-08 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypercholesterolemia
Keywords: LDL, HDL
MeSH Terms: conditions — Hypercholesterolemia | interventions — pitavastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pitavastatin 4mg (Active Comparator): Pitavastatin 4mg tablet by mouth once daily for 12 weeks
  Interventions: Drug: Atorvastatin 20mg; Drug: Rosuvastatin 5mg
- Atorvastatin 20mg (Active Comparator): Atorvastatin 20mg tablet by mouth once daily for 12 weeks
  Interventions: Drug: Pitavastin 4mg; Drug: Rosuvastatin 5mg
- rosuvastatin 5 mg (Active Comparator): rosuvastatin 5 mg tablet by mouth once daily for 12 weeks
  Interventions: Drug: Pitavastin 4mg; Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Pitavastin 4mg
  Other Names: Livalo
  Arms: Atorvastatin 20mg; rosuvastatin 5 mg
Drug: Atorvastatin 20mg
  Other Names: Lipitor
  Arms: Pitavastatin 4mg; rosuvastatin 5 mg
Drug: Rosuvastatin 5mg
  Other Names: Crestor
  Arms: Atorvastatin 20mg; Pitavastatin 4mg

SUMMARY:
The purpose of this study is to determine if Pitavastatin lowers CoQ10 less than Atorvastatin or Rosuvastatin.

DETAILED DESCRIPTION:
Statins are known effectively treat high cholesterol and heart disease. However, statins may lower endogenous levels of Coenzyme10 (CoQ10). This decrease in CoQ10 levels may be responsible for side effects such as myalgia.

Previous studies have shown that Pitavastatin may not affect CoQ10 levels as other statins do, while still lowering cholesterol.

In this study, investigators intend to compare the plasma levels of CoQ10 in patients taking 3 different FDA-approved statins, in equipotent doses.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C levels of 100-200mg/dl; triglycerides </=200mg/dl at screening visit
* Willing to discontinue use of all lipid-altering doses fo medication or supplements for the duration of the study

Exclusion Criteria:

* LDL-C <100mg/dl or >200mg/dl, Triglycerides >200mg/dl
* History of diabetes mellitus or documented fasting blood glucose >125mg/dl or HbA1c >6.4%
* History of coronary artery disease
* history of chronic renal or hepatic disease
* known sensitivity of intolerance to a statin
* persistent elevated liver enzymes or CPK (>3 x upper normal limit)
* currently taking CoQ10 supplements and unable discontinue for duration of study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Moriarty, MD, FACC, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin 20mg: Atorvastatin 20mg, once daily by mouth for 12 weeks
- Pitavastatin 4mg: Pitavastatin 4mg, once daily by mouth for 12 weeks
- Rosuvastatin 5 mg: Rosuvastatin 5mg, once daily by mouth for 12 weeks
Period: Enrollment and Washout
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Started | 45 | 45 | 44
Completed | 45 | 45 | 44
Not Completed | 0 | 0 | 0
Period: Randomization
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Started | 45 | 45 | 44
Completed | 45 | 45 | 44
Not Completed | 0 | 0 | 0
Period: End of Treatment
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Started | 45 | 45 | 44
Completed | 44 | 39 | 43
Not Completed | 1 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg | Total
Number analyzed (Participants) | 45 | 45 | 44 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.68 (12.52) | 56.66 (9.93) | 56.08 (12.28) | 55.80 (11.57)
Gender [Count of Participants; unit: Participants]
  Female | 28 | 30 | 36 | 94
  Male | 17 | 15 | 8 | 40
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 44 | 134
Waist Size [Mean (Standard Deviation); unit: inches] | 36.41 (5.76) | 37.45 (4.20) | 34.54 (5.60) | 36.12 (5.33)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Plasma CoQ10 Levels
Description: Change in levels will be measured by taking difference between Baseline and Week 12 measures.
Time Frame: Change from Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 42 | 40 | 36
μg/g
  Ubiquinone | -96.70 (224.24) | -110.42 (136.29) | -103.91 (237.27)
  Total CoQ10 | -721.09 (830.47) | -464.85 (571.37) | -642.43 (874.99)
  Upiquinol | -624.39 (669.45) | -354.43 (544.42) | -538.52 (709.53)

2. Secondary Outcome: Changes in Major Lipid Parameters - VLDL Size
Description: Change in levels will be measured by difference in levels at 12 weeks. Measure based on VLDL size.
Time Frame: Change from Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: nanometre (nm)
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 44 | 43 | 37
nanometre (nm) | 0.68 (5.63) | 0.81 (5.84) | 3.17 (6.25)

3. Secondary Outcome: Changes to Glucose Metabolism - HbA1c and Insulin
Description: Change in levels will be measured by levels at 12 weeks minus levels at baseline. Changes measured based in HbA1c, and insulin.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change from baseline measure
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 44 | 42 | 37
percentage change from baseline measure
  HbA1c | 0.00 (0.03) | 0.00 (0.04) | 0.00 (0.04)
  Insulin | 0.16 (0.47) | 0.01 (0.43) | 0.17 (0.38)

4. Secondary Outcome: Changes in HDL and LDL Size
Description: Change in levels will be measured by difference in levels at 12 weeks
Time Frame: Change from Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: nanometre (nm)
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 42 | 43 | 36
nanometre (nm)
  HDL Size | 0.23 (0.27) | 0.23 (0.26) | 0.12 (0.32)
  LDL Size | -0.02 (0.44) | -0.11 (0.43) | -0.09 (0.41)

5. Secondary Outcome: Changes to Glucose Metabolism - Fructosamine
Description: Change in levels will be measured by levels at 12 weeks minus levels at baseline. Changes measured based in fructosamine.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: µmol
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 33 | 30 | 27
µmol | 1.91 (17.16) | -1.17 (13.74) | -3.07 (14.77)

6. Secondary Outcome: Changes HDL Particle Number and LDL Particle Number
Description: Change in levels will be measured by difference in levels at 12 weeks.
Time Frame: Change from Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: particle number
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Number analyzed (Participants) | 42 | 43 | 36
particle number
  HDL Particle Number | 0.64 (5.24) | 2.55 (4.19) | 2.05 (5.17)
  LDL Particle Number | -873.48 (353.76) | -768.26 (334.01) | -626.61 (341.28)

ADVERSE EVENTS:
Arm/Group | Atorvastatin 20mg | Pitavastatin 4mg | Rosuvastatin 5 mg
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 1/45 | 2/45 | 5/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 20mg (N=45) | Pitavastatin 4mg (N=45) | Rosuvastatin 5 mg (N=44)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes